CLINICAL TRIAL: NCT05798728
Title: Outpatient Transcervical Balloon: Does it Shorten the Hospital Stay for Induction of Labor? Randomized Control Trial
Brief Title: Outpatient Transcervical Balloon For Induction of Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hurley Medical Center (Other)
Responsible Party: Principal Investigator, Atinuke Akinpeloye, Core faculty in the department of Obstetrics and Gynecology, Hurley Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1914347
Record Dates: First submitted 2023-03-07; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Induced Vaginal Delivery; Induced; Birth
Keywords: Misoprostol; Cytotec; Cervical ripening; Outpatient; Inpatient; Transcervical foley balloon; Mechanical dilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpatient Vaginal Misoprostol (Active Comparator): These participants will receive intravaginal Misoprostol in the inpatient setting per our standard hospital protocol for cervical ripening.
  Interventions: Procedure: Inpatient Vaginal Misoprostol
- Outpatient transcervical foley balloon (Experimental): These participants will receive a catheter which will be placed by a physician present in the clinic, however, patient are discharged home for 12 hours until their time of induction of labor.
  Interventions: Procedure: Outpatient transcervical foley balloon

INTERVENTIONS:
Procedure: Outpatient transcervical foley balloon — These participants will receive a 16-French Foley catheter which will be placed by a physician present in the clinic. The balloon will be inflated with 40 mL of sterile water, and the catheter will then be gently withdrawn so that the balloon applies pressure against the internal os. The catheter will then be taped to the inner thigh.
  Arms: Outpatient transcervical foley balloon
Procedure: Inpatient Vaginal Misoprostol — These participants will receive 25 micrograms of Misoprostol (100- microgram tablet cut into fourths by the hospital pharmacist) inserted vaginally into the posterior fornix every 4 hours and repeated up to a maximum of six doses per our standard hospital protocol.
  Arms: Inpatient Vaginal Misoprostol

SUMMARY:
The goal of this randomized control trial is to compare outpatient transcervical foley balloon to inpatient vaginal misoprostol in pregnant women for cervical ripening. The main questions it aims to answer are:

1. Does outpatient transcervical foley balloon decreased the time from admission to delivery compared to inpatient vaginal misoprostol
2. Does outpatient transcervical foley balloon will increase risk of c-section during induction of labor compared to inpatient vaginal misoprostol

Participants will be randomized to either the outpatient transcervical foley balloon group or to the inpatient intravaginal misoprostol group. The researchers will compare if outpatient transcervical foley balloon decreases the tie from hospital admission to delivery of the baby.

DETAILED DESCRIPTION:
This is a prospective randomized unblinded control trial. Consented patients will have a cervical exam performed in the clinic to confirm that the bishop score is less than 6. Once this and the inclusion criteria are met, the participant will be randomized to either the outpatient transcervical foley arm or the vaginal misoprostol arm. Each pregnant woman will undergo the intervention stated in the numbered envelope which will be distributed based on their order of inclusion in the study. Due to the nature of the procedure, blinding could not be done.

Participants randomized to the transcervical foley group will be scheduled an appointment in the clinic the day before their scheduled induction day for the final screen and foley placement. On the other hand, participants randomized to the vaginal misoprostol group will be admitted to the labor and delivery unit on the day of their scheduled induction. All participants will undergo a cervical examination before the assigned intervention to verify their eligibility status. Those who do not meet the eligibility criteria, will be excluded. Both transcervical foley and vaginal misoprostol are standard of care for induction of labor at Hurley Medical Center. Thus, there would be no additional cost to the patient. The only difference in the study is the setting in which the transcervical foley is placed, i.e. in the obstetrics clinic as an outpatient.

Oxytocin will be initiated in all patients who did not have at least three regular contractions in 10 minutes. Continuous fetal heart rate monitoring and uterine activity monitoring will be performed in all patients. Amniotomy will be performed during the course of labor at the discretion of the health care provider and epidural anesthesia will be administered per the patient's request.

ELIGIBILITY:
Inclusion Criteria:

1. Term singleton pregnancy (37 weeks of gestation or greater)
2. Bishop score less than 6 and a maximum cervical dilation of 2 cm
3. Cephalic presentation

Exclusion Criteria:

1. Rupture of membranes
2. Regular uterine contractions (3 or more contractions per 10 minutes)
3. History of prior uterine surgery (cesarean delivery or myomectomy)
4. Multiples gestations
5. Malpresentation
6. Nonreassuring fetal heart tracing (category 3 or persistent category 2)
7. Fetal demise
8. Anomalous fetus
9. Any contraindication to vaginal delivery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-06-09 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Time from hospital admission to delivery of the newborn | From hospital admission until delivery of the newborn
  The primary outcome is to determine if there is a difference in the time from admission to delivery for those who receive transcervical foley balloon in the clinic the day before induction compared to those who get vaginal misoprostol in the hospital on the day of the induction

SECONDARY OUTCOMES:
Chorioamnionitis/endometritis | From hospital admission until 2 weeks postpartum
  Number of participants with fever, increased white blood cell count or foul smelling discharge in the outpatient transcervical foley group compared to that of in the intravaginal Misoprostol group
Cesarean delivery | From hospital admission until delivery of the newborn
  Number of participants delivering via cesarean section in the outpatient transcervical foley group compared to that of in the inpatient intravaginal Misoprostol group
Postpartum hemorrhage | From hospital admission until 2 weeks postpartum
  Number of participants with quantified blood loss greater than 1000ml in the outpatient transcervical foley group compared to that of in the inpatient intravaginal Misoprostol group
Delivery within 24 hours of hospital admission | From hospital admission until delivery of the newborn
  To determine is if the delivery rate within 24 hours from hospital admission in the outpatient transcervical foley group is greater compared to the inpatient intravaginal Misoprostol group
Total hospital length of stay | From hospital admission until discharge, assessed up to a week
  To determine is if there is an increase risk of prolonged hospital stay in the outpatient transcervical foley group compared to the inpatient intravaginal Misoprostol group
Hospital readmission within 30 days of discharge | From discharge until 30 days postpartum
  To determine is if there is an increase risk of hospital readmission within 30 days of discharge in the outpatient transcervical foley group compared to the inpatient intravaginal Misoprostol group
Cervical examination at the time of admission | Within the first hour of hospital admission
  To determine if cervical dilation is more favorable for induction in the outpatient transcervical foley balloon compared to the inpatient intravaginal Misoprostol
Unscheduled hospital admissions or unscheduled visits to our obstetric triage unit before the time of scheduled admission | From date of outpatient transcervical foley balloon placement until time of scheduled admission, assessed up to 12 hours
  To determine if outpatient transcervical foley balloon placement increases the unscheduled hospital admissions or unscheduled visits to our obstetric triage unit before the time of scheduled admission.
Frequency of acetaminophen use after randomization but before hospital admission | From time of outpatient transcervical foley balloon placement until hospital admission, assessed up to 12 hours
  To determine if outpatient transcervical foley balloon placement increases the frequency of acetaminophen use after randomization but before hospital admission
Spontaneous rupture of membranes between randomization and hospital admission | From time of transcervical foley balloon placement until spontaneous rupture of membranes, assessed up to 12 hours
  To determine if outpatient transcervical foley balloon placement increases spontaneous rupture of membranes between randomization and hospital admission
Duration of oxytocin infusion (in min) | From hospital admission until delivery of the newborn
  To determine if there is an increase in the duration of oxytocin infusion (in minutes) in the outpatient transcervical foley group compared to the inpatient intravaginal Misoprostol group
Maximum oxytocin rate infused (in milliunits/min) | From hospital admission until delivery of the newborn
  To determine if there is an increase in the maximum oxytocin rate infused (in milliunits/min) in the outpatient transcervical foley group compared to the inpatient intravaginal Misoprostol group
Duration of neuraxial anesthesia use | From hospital admission until delivery of the newborn
  To determine is if there is an increase in the duration of neuraxial anesthesia use in the outpatient transcervical foley group compared to the inpatient intravaginal Misoprostol group
Presence of heavy vaginal bleeding before delivery | From outpatient transcervical foley balloon insertion until delivery of newborn
  To determine if outpatient transcervical foley balloon placement increases heavy vaginal bleeding before delivery
Meconium-stained amniotic fluid | From hospital admission until delivery of the newborn
  To determine is if there is an increase in the rate of meconium-stained amniotic fluid in the outpatient transcervical foley group compared to the inpatient intravaginal Misoprostol group
Time from rupture of membranes to delivery | From time of rupture of membranes until delivery of the newborn
  To determine is if there is an decreases the duration from rupture of membranes to delivery in the outpatient transcervical foley group compared to the inpatient intravaginal Misoprostol group
Highest maternal intrapartum temperature | From hospital admission until delivery of the newborn
  To determine is if there is an increase in maternal intrapartum temperature in the outpatient transcervical foley group compared to the inpatient intravaginal Misoprostol group
Admission white blood cell count | From hospital admission until delivery of the newborn
  To determine is if there is an increase in admission white blood cell count in the outpatient transcervical foley group compared to the inpatient intravaginal Misoprostol group

CONTACTS AND LOCATIONS:
Overall Officials: Atinuke Akinpeloye, MD, Principal Investigator — Hurley Medical Canter
Locations (1):
- Hurley Medical Center, Flint, Michigan, United States